CLINICAL TRIAL: NCT02564874
Title: Effect on Dietary Compensation and Weight Gain in Adults by Savory Solid and Sugary Liquid Discretionary Food Sources
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1505M71543
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain

ARMS (2):
- Savory snack (Experimental): 1-2 assigned snacks to be taken in determined portions equivalent to 15% of dietary energy intake, chosen from 9-point hedonic preferences questionnaire completed by participant (chips, pretzels, etc.)
  Interventions: Other: Discretionary calorie source
- Sugary beverage (Experimental): 1-2 soda-based drinks/juice to be taken in determined portions equivalent to 15% of dietary energy intake, chosen from 9-point hedonic preferences questionnaire completed by participant (coke, sprite, etc.)
  Interventions: Other: Discretionary calorie source

INTERVENTIONS:
Other: Discretionary calorie source — We are assigning participants randomly to either of two different sources of discretionary calories (savory snacks or sugary beverages)

SUMMARY:
The objective of this study is to determine the effect different sources and forms of discretionary foods have on dietary compensation and energy intake in healthy adults in a free living, real world setting. Specifically, this pilot study will compare the effect of the greatest caloric sources of savory and sweetened discretionary foods in the American diet (savory snacks v. sugar-sweetened beverages). The rationale for conducting this study is to test the mechanism whereby sugar-sweetened beverages are hypothesized to relate to weight gain and obesity above and beyond other discretionary foods (lack of energy intake compensation due to liquid form of the beverage), since the evidence for this topic is limited. The subject population will be 20 men and women between the age of 18 and 59 who are overweight by body mass index (BMI ≥ 25 kg/m2), generally healthy, consume sugar-sweetened beverages or , and are willing to incorporate a sweetened beverage or a savory snack into their usual diet in the 4 week period.

DETAILED DESCRIPTION:
The study design will be a randomized parallel study consisting of a 4-week period during which each participant will be assigned to one of the two food groups. Participants in each group will be provided with a daily provision of a chosen sugar-sweetened beverage or savory snack to incorporate into their usual dietary pattern. The main outcome is dietary intake, specifically energy intake gathered by 24 hour dietary recalls. Secondary outcomes include measured body weight / BMI. The participant will be blinded to the main outcome so as not to affect the results. To do this they will be told the rationale for the study is to examine the effect of discretionary food sources on perceived health status and provided a standard, valid short questionnaire (SF-12) at the beginning, middle and end of each period. Investigators will estimate the energy intake necessary for weight maintenance of the subject based upon a standard approach and equation that accounts for the participant's age, sex, body size, and activity level. The subject will be provided with approximately 15-20% of their estimated daily energy needs in the form of a sugar-sweetened beverage or savory snack of their choice during one period and will be asked to incorporate this into their usual dietary pattern each day for 4 weeks. During the 4 week period the subject will be randomly prompted to complete five, 24-hour dietary recalls using an online tool. They will also be asked to fill out a short physical activity questionnaire during the intervention periods and a short questionnaire on perceived health (SF-12). They will have their weight, height, and waist circumference measured at the beginning and end of the period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* overweight (BMI ≥ 25 kg/m2)
* consume sugar-sweetened beverages or savory snacks
* willing to consume amount of beverages and food provided to supplement usual dietary habits during the study period

Exclusion Criteria:

* Recently lost a significant amount of weight or looking to lose weight
* recently begun a new diet or exercise regimen
* prevalent or history of major illnesses or chronic disease (e.g. diabetes, heart disease, cancer, other metabolic disorders) which may affect adherence
* pregnant
* use of prescription medications (aside from birth control)
* report ≥ 1 alcoholic beverage a day
* currently smoke
* report being a restrained eater or having < 51% of control over the selection and preparation of the food they eat
* adults lacking capacity to consent for self

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Dietary energy compensation as measured by weight changes | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- West Bank Office Building, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Almiron-Roig E, Palla L, Guest K, Ricchiuti C, Vint N, Jebb SA, Drewnowski A. Factors that determine energy compensation: a systematic review of preload studies. Nutr Rev. 2013 Jul;71(7):458-73. doi: 10.1111/nure.12048. Epub 2013 Jun 10. PMID 23815144
- [Background] Popkin BM, Armstrong LE, Bray GM, Caballero B, Frei B, Willett WC. A new proposed guidance system for beverage consumption in the United States. Am J Clin Nutr. 2006 Mar;83(3):529-42. doi: 10.1093/ajcn.83.3.529. PMID 16522898
- [Background] Little TJ, Feinle-Bisset C. Effects of dietary fat on appetite and energy intake in health and obesity--oral and gastrointestinal sensory contributions. Physiol Behav. 2011 Sep 26;104(4):613-20. doi: 10.1016/j.physbeh.2011.04.038. Epub 2011 May 3. PMID 21596051
- [Background] Pereira, Mark A. The possible role of sugar-sweetened beverages in obesity etiology: a review of the evidence. Int J Obes. 2006. 30. 28-36.
- [Background] USDA Dietary Guidelines Advisory Committee. (2005). Discretionary calories. In The Report of the Dietary Guidelines Advisory Committee on Dietary Guidelines for Americans, 2005(6th ed.). United States Department of Agriculture.